CLINICAL TRIAL: NCT00734643
Title: Family Stress, Coping and Outcomes Following the Diagnosis of Hypoplastic Left Heart Syndrome in a Newborn
Brief Title: Family Adaptation Study Following the Diagnosis of Hypoplastic Left Heart Syndrome in a Newborn
Status: Completed | Type: Observational
Sponsor: Medical College of Wisconsin (Other)
Collaborators: Children's Hospital and Health System Foundation, Wisconsin (Other); American Nurses Foundation (Other); Columbia University (Other); Boston Children's Hospital (Other); University of Michigan (Other); Children's Hospital of Philadelphia (Other); Johns Hopkins All Children's Hospital (Other); Medical University of South Carolina (Other); Arkansas Children's Hospital Research Institute (Other); Nicklaus Children's Hospital f/k/a Miami Children's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CHW 06/117
Record Dates: First submitted 2008-08-13; First posted 2008-08-14 (Estimated); Last update posted 2020-01-29 (Actual); Status verified 2020-01

CONDITIONS: Hypoplastic Left Heart Syndrome
Keywords: Hypoplastic Left Heart Syndrome; Family coping; Complex Congenital Heart Disease
MeSH Terms: conditions — Hypoplastic Left Heart Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Survival for one of the most complex forms of congenital heart disease, hypoplastic left heart syndrome (HLHS), has improved dramatically. However, little is known about family stress, coping and outcomes following the diagnosis of HLHS. It is expected that families face emotional, social and financial stressors. Health care professionals have a unique opportunity to positively influence how families interpret and adapt to these stressors. The specific aims of the study are to describe perceived stress, and coping skills utilized, in parents of children with HLHS and their impact on family outcomes measured as well-being, adaptation and caregiver/family quality of life, and to describe changes in stress, coping, and adaptation and differences in perceptions of mothers versus fathers of children with HLHS over the first 14 months of life. The Resiliency Model of Family Adjustment and Adaptation (McCubbin, Thompson, & McCubbin, 1996) is the theoretical framework that guides this research.

Hypotheses:

1. Family perception of stress, and coping skills utilized, will have an impact on family outcomes measured as well-being, adaptation, and caregiver/family quality of life.
2. Variables influencing perception of stress and variables influencing family coping will be significant predictors of family adaptation outcomes.
3. Perceptions of stress, coping skills utilized, and family adaptation outcomes will improve during the first 14 months of life with an infant with HLHS.
4. Mothers and fathers will report different perceptions of stress, coping skills utilized, and family adaptation outcomes during the first 14 months of life with an infant with HLHS.

ELIGIBILITY:
Inclusion Criteria:

* Parents of all patients diagnosed with complex congenital heart disease requiring hospitalization or intervention during the neonatal period

Exclusion Criteria:

* Parents unable to speak or read English

Max Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Parents of all patients diagnosed with complex congenital heart disease requiring hospitalization or intervention during the neonatal period will be eligible to participate. Parents unable to speak or read English will be excluded. An attempt will be made to obtain consent for participation from both the mother and father of the affected infant. If no father is involved in the care of the infant, measures will be obtained from mothers alone. The model will be tested using mothers' reports of family variables. Single parents will be able to participate but will not be included in comparisons between mothers and fathers. Nurse coordinators at participating centers will conduct subject screening and consenting.
Sampling Method: Non-Probability Sample
Enrollment: 213 (Actual)
Dates: Start 2006-06; Primary Completion 2011-05 (Actual); Study Completion 2019-09-05 (Actual)

PRIMARY OUTCOMES:
Family Adaptation | 14 months
  Family adaptation will be measured with the general functioning scale of the Family Assessment Device (FAD) (Miller, Epstein, Bishop & Keitner, 1985) at T1, T2 and T3. The FAD provides an overall measure of family functioning; 12 items, reliability alpha = .83-.86.

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen A Mussatto, PhD, RN, Principal Investigator — Children's Hospital and Health System Foundation, Wisconsin
Locations (1):
- Children's Hospital of Wisconsin, Milwaukee, Wisconsin, United States